CLINICAL TRIAL: NCT04969029
Title: Randomized, Controlled Phase II Study of Immunotherapy Versus Standard Chemotherapy as Adjuvant Therapy After Surgery for Colon Cancer With MSI-H or POLE/ POLD1 Mutations
Brief Title: Immunotherapy Versus Chemotherapy as Adjuvant Therapy for Colon Cancer With MSI-H or POLE/ POLD1 Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJMUCH-GI-CRC01
Record Dates: First submitted 2021-07-05; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Immunotherapy; Adjuvant Therapy; Colon Cancer; MSI-H
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immunotherapy (Experimental): In the immunotherapy group, the treatment regimen was Tirelizumab 200mg, intravenously infused once every 3 weeks until the end of 12 months of treatment, with a total of 17 infused times.
  Interventions: Drug: Tirelizumab
- chemotherapy (No Intervention): The chemotherapy regimen of the standard chemotherapy group was XELOX regimen, oxaliplatin 130mg/m2, d1, capecitabine 1000mg/m2, orally, bid (half an hour after breakfast and dinner), d1-14, every 21 days. The duration of treatment was determined according to the patient's postoperative pathological stage (3 months for T4N0/ T1-3N1 and 6 months for T4N+/ T1-3N2).

INTERVENTIONS:
Drug: Tirelizumab — In the immunotherapy group, the treatment regimen was Tirelizumab 200mg, intravenously infused once every 3 weeks until the end of 12 months of treatment, with a total of 17 infused times.
  Arms: immunotherapy

SUMMARY:
This is a two-group, parallel, randomized, standard-control phase II study comparing the safety and efficacy of immunotherapy versus standard chemotherapy in patients undergoing T4NX/TXN+ colon cancer surgery with MSI-H or POLE/ POLD1 mutations.This study was conducted in the Department of Gastroenterology, Tumor Hospital of Tianjin Medical University.

Patients with MSI-H or POLE/ POLD1 gene mutations confirmed by PCR sequencing or NGS sequencing will be randomly assigned (2:1) to immunotherapy (experimental group) or standard chemotherapy (control group) after signing informed consent. In this study, 30 patients will be enrolled, 20 patients will receive immunotherapy and 10 patients will receive standard chemotherapy.

In the immunotherapy group, the treatment regimen was Tirelizumab 200mg, intravenously infused once every 3 weeks until the end of 12 months of treatment, with a total of 17 infused times. Patients enrolled in this group could enjoy the preferential policy of purchasing 7 times and giving 10 times at their own expense.

The chemotherapy regimen of the standard chemotherapy group was XELOX regimen, oxaliplatin 130mg/m2, d1, capecitabine 1000mg/m2, orally, bid (half an hour after breakfast and dinner), d1-14, every 21 days. The duration of treatment was determined according to the patient's postoperative pathological stage (3 months for T4N0/ T1-3N1 and 6 months for T4N+/ T1-3N2).

Patients received regular and periodic reviews, with imaging evaluations every 3 months for the first 2 years and every 6 months after 2 years. Safety will be evaluated by AE and laboratory tests. After tumor recurrence or metastasis was first detected, tumor tissue biopsies were taken again for NGS sequencing, and all patients were followed up every 3 months until death according to the plan.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent.
2. Age ≥18.
3. Colonic adenocarcinoma confirmed histologically or histopathologically.
4. No residual cancer was confirmed after radical resection of colon cancer.
5. According to the overall postoperative results, T4NX/TXN+ colon cancer was determined according to AJCC/ UICC TNM staging eighth edition.
6. No liver, peritoneum or other distant metastases.
7. MSI-H or POLE/ POLD1 gene mutation was confirmed by PRC or NGS sequencing.
8. ECOG physical status score is 0 or 1.
9. Appropriate organ function according to the following laboratory test values obtained within 7 days prior to use on Day 1 of Cycle 1:

   A. Hemoglobin value ≥9.0g/dL. B. Absolute neutrophil count ≥1,500/mm3 (≥1.5*109/L). C. Platelet count ≥100,000/mm3 (≥100*109/L). D. Total serum bilirubin ≤1.5* upper normal limit (ULN). E. aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5* upper limit of normal value (ULN).

   F. Serum creatinine ≤1.5 times * upper limit of normal (ULN) or creatinine clearance ≥50ml/min.
10. Willing and able to follow research procedures and visit plans.

Exclusion Criteria:

1. The patient had received non-surgical treatment for colon cancer (e.g., radiation, chemotherapy, and hormone therapy).
2. Has a serious illness or medical condition, including but not limited to the following:

   A. Recurrent in situ or metastatic tumor of any other site is known. B. Systemic active infection (i.e., infection causes body temperature ≥38℃). C. Clinically significant intestinal obstruction, pulmonary fibrosis, renal failure, liver failure, or symptomatic cerebrovascular disease.

   D. Severe/unstable angina, New York Heart Association (NYHA) grade III or IV symptomatic congestive heart failure.

   E. Gastrointestinal bleeding of clinical significance. F. Known presence of human immunodeficiency virus (HIV) or acquired routine immunodeficiency syndrome (AIDS) -associated disease, or active hepatitis B or C.
3. Pregnant or lactating women.
4. The researcher did not consider it appropriate to enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
3-year relapse-free survival | 60 months
  The time from the beginning of randomization to the time when the disease recurs or the patient dies from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No